CLINICAL TRIAL: NCT05314582
Title: Investigation of the Effects of Anticoagulant/Antiaggregant Use on Postoperative Bleeding Risk in Patients Operated for Bladder Tumor and Benign Prostatic Hyperplasia
Brief Title: Anticoagulant/Antiaggregant Use and Postoperative Bleeding Risk in Patients With Bladder Tumor and Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Abdullah İlktaç, Pincipal investigator, Bezmialem Vakif University
Other Study IDs: 196083
Record Dates: First submitted 2022-03-27; First posted 2022-04-06 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Hematuria; Retention, Urinary; Operative Bleeding; Blood Transfusion Complication
Keywords: bladder cancer; benign prostatic hyperplasia; transurethral resection; hematuria
MeSH Terms: conditions — Hematuria; Urinary Retention; Transfusion Reaction; Urinary Bladder Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- TURP patients using anticoagulant/antiaggregant medication: Patients who used anticoagulant/antiaggregant medication for any reason (eg: coronary artery disease, atrial fibrillation, cerebrovascular disease) before surgery and underwent endoscopic prostatectomy (TURP).
- TURP patients not using anticoagulant/antiaggregant medication: Patients with no history of anticoagulant/antiaggregant medication and underwent endoscopic prostatectomy (TURP).
- TUR-BT patients using anticoagulant/antiaggregant medication: Patients who used anticoagulant/antiaggregant medication for any reason (eg: coronary artery disease, atrial fibrillation, cerebrovascular disease) before surgery and underwent endoscopic bladder tumor resection (TUR-BT).
- TUR-BT patients not using anticoagulant/antiaggregant medication: Patients with no history of anticoagulant/antiaggregant medication and underwent endoscopic bladder tumor resection (TUR-BT).
- Open prostatectomy patients using anticoagulant/antiaggregant medication: Patients who used anticoagulant/antiaggregant medication for any reason (eg: coronary artery disease, atrial fibrillation, cerebrovascular disease) before surgery and underwent open prostatectomy (OP).
- Open prostatectomy patients not using anticoagulant/antiaggregant medication: Patients with no history of anticoagulant/antiaggregant medication and underwent open prostatectomy (OP).

SUMMARY:
Patients who were using anticoagulant or antiaggregant medications for any reason and underwent transurethral resection of bladder tumor (TUR-BT) or transurethral resection of the prostate (TURP) or open prostatectomy (OP) due to BPH will be compared with those who were not using anticoagulant or antiplatelet medication. The rates of postoperative clot retention, presence of hematuria, reoperation due to hematuria, blood transfusion and re-admissions due to hematuria in the first postoperative month will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing complete endoscopic transurethral tumor resection (TUR-BT) for bladder cancer
* Patients undergoing TURP due to benign prostatic hyperplasia
* Patients undergoing open prostatectomy due to benign prostatic hyperplasia

Exclusion Criteria:

* Patients who underwent incomplete transurethral tumor resection for bladder cancer
* Patient who underwent TUR biopsy for restaging with no obvious macroscopic tumoral lesion
* Patients who underwent cystectomy for bladder cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were referred to endoscopic bladder tumor resection (TUR-BT) or open or endoscopic BPH surgery (TURP or open prostatectomy) will be included in this study. For patients using anticoagulant/antiaggregant medications, relevant specialty (eg: Cardiology, neurology, cardiovascular surgery) or anesthesiologist will decide whether the patient will quit these medications before surgery or not, when to quit and whether low molecular weight heparin will be started instead. The responsible physician of the patient will decide when to restart the anticoagulant therapy after the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Episode of clot retention | Immediately after the surgery up to 1 month
  Presence of clot retention due to hematuria after the operation which requires manuel irrigation
Requirement of blood transfusion | Immediately after the surgery up to 1 month
  Gross hematuria requiring blood transfusion
Re-operation rates | Immediately after the surgery up to 1 month
  Re-operation requirement for hematuria
Duration of hospitalization | Immediately after the surgery up to discharge
  Duration of hospitalization
Rate of re-admission | From discharge up to one month
  Rate of re-admission due to hematuria

SECONDARY OUTCOMES:
Postoperative hematocrit/hemoglobin levels | Immediately after the surgery up to discharge
  Change in the Postoperative hematocrit/hemoglobin levels compared to the preoperative values.
Amount of irrigation volume | Immediately after the surgery up to discharge
  Amount of postoperative continuous bladder irrigation volume

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Ilktac, MD, Study Chair — Bezmialem Vakif University, Faculty of Medicine, Department of Urology
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)